CLINICAL TRIAL: NCT05383989
Title: UniVenture: A Partnership to Address Heavy Drinking and Other Substance Misuse on Canadian University Campuses
Brief Title: The UniVenture Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherry Stewart (Other)
Collaborators: Dalhousie University (Other); St. Francis Xavier University (Unknown); Université de Montréal (Other); York University (Other); University of British Columbia (Other); University of Victoria (Other); Canadian Centre on Substance Use and Addiction (CCSA) (Unknown); Canadian Research Initiative in Substance Misuse (Other); Injury Free Nova Scotia (IFNS) (Unknown); Mental Health Commission of Canada (MHCC) (Unknown); Postsecondary Education Partnership - Alcohol Harms (PEP-AH) (Unknown); Strategy for Patient Orientated Research (Unknown); SHARP- Students for Healthy Alternatives & Risk Prevention (Unknown); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Sherry Stewart, Professor, Dalhousie University
Organization: Dalhousie University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-5689
Record Dates: First submitted 2021-09-27; First posted 2022-05-20 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Anxiety Sensitivity; Hopelessness; Sensation Seeking; Impulsivity
Keywords: Substance misuse; Prevention; Personality; Knowledge mobilization; Well-being; Academic retention; Academic performance; Binge drinking; Emerging adulthood; Life transitions; Technology assisted programs; Student services
MeSH Terms: conditions — Impulsive Behavior; Binge Drinking

STUDY DESIGN:
Intervention Model Description: 1. A personality-matched wellness program condition in face-to-face format (i.e., high AS student receives face-to-face AS program; high HOP student receives face-to-face HOP workshop: high SS student receives face-to-face SS workshop; high IMP student receives face-to-face IMP workshop)
  2. A personality-matched wellness program condition in distance-delivery format (i.e., high AS student receives distance-delivered AS workshop; etc. as per the face-to-face format).
  3. Services-as-usual offered by the respective university
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UniVenture- face-to-face (in-person format) (Experimental): Personality-matched wellness program condition in face-to-face format (i.e., high AS student receives face-to-face AS program; high HOP student receives face-to-face HOP workshop: high SS student receives face-to-face SS workshop; high IMP student receives face-to-face IMP workshop)
  Interventions: Behavioral: UniVenture Hopelessness manual; Behavioral: UniVenture Anxiety Sensitivity manual; Behavioral: UniVenture Sensation Seeking manual; Behavioral: UniVenture Impulsivity manual
- UniVenture- online (distance-delivery format) (Active Comparator): Personality-matched wellness program condition in distance-delivery format (i.e., high AS student receives online (distance-delivered) AS workshop; high HOP student receives online (distance-delivered) HOP workshop: high SS student receives online (distance-delivered) SS workshop; high IMP student receives online (distance-delivered) IMP workshop
  Interventions: Behavioral: UniVenture Hopelessness manual; Behavioral: UniVenture Anxiety Sensitivity manual; Behavioral: UniVenture Sensation Seeking manual; Behavioral: UniVenture Impulsivity manual
- UniVenture- service as usual (control) (Placebo Comparator): Services-as-usual offered by the respective university
  Interventions: Behavioral: Service as usual provided by the University

INTERVENTIONS:
Behavioral: UniVenture Hopelessness manual — Intended for those who score at least 0.5 standard deviation (SD) above the population-specific norm on Hopelessness (HOP) personality traits on the Substance Use Risk Profile Scale (SURPS).
  Arms: UniVenture- face-to-face (in-person format); UniVenture- online (distance-delivery format)
Behavioral: UniVenture Anxiety Sensitivity manual — Intended for those who score at least 0.5 standard deviation (SD) above the population-specific norm on Anxiety Sensitivity (AS) personality traits on the Substance Use Risk Profile Scale (SURPS).
  Arms: UniVenture- face-to-face (in-person format); UniVenture- online (distance-delivery format)
Behavioral: UniVenture Sensation Seeking manual — Intended for those who score at least 0.5 standard deviation (SD) above the population-specific norm on Sensation Seeking (SS) personality traits on the Substance Use Risk Profile Scale (SURPS)
  Arms: UniVenture- face-to-face (in-person format); UniVenture- online (distance-delivery format)
Behavioral: UniVenture Impulsivity manual — Intended for those who score at least 0.5 standard deviation (SD) above the population-specific norm on Impulsivity (IMP) personality traits on the Substance Use Risk Profile Scale (SURPS).
  Arms: UniVenture- face-to-face (in-person format); UniVenture- online (distance-delivery format)
Behavioral: Service as usual provided by the University — It is the regular university-provided well-being services.
  Arms: UniVenture- service as usual (control)

SUMMARY:
UniVenture is a research partnership with one common goal: to adapt, test, and begin sharing an effective, sustainable, targeted wellness program to tackle the timely social issue of heavy drinking and other substance misuse on Canadian campuses. Our project is a 5-year, multi-site, controlled study involving 1st and 2nd year undergraduates at 5 representatively diverse Canadian university sites (Dalhousie University, St. Francis Xavier University, York University, Université de Montréal, and University of British Columbia-Okanagan). The investigator will test a program targeting personality traits linked to substance misuse. An earlier version of this program led to marked reductions in substance use and distress in adolescents. Our novel objectives are to examine the program's effects on substance use and distress among emerging adults; uptake of prescription drug use given the opioid crisis; and undergraduates' academic success. The investigator will carry out a randomized controlled trail in which two versions of the program will be assessed: a face-to-face and an innovative and accessible technology-assisted distance-delivery format, both compared to normal campus services alone. UniVenture may potentially have a dramatic effect on university policies on the prevention of substance misuse on Canadian campuses by helping partners appreciate the effectiveness of targeted and personalized approaches, and leveraging partners' expansive networks to inform other Canadian universities. A successful technology-assisted distance-delivered program will provide universities with an effective, relatively low-cost, and accessible tool to intervene with risky substance use behaviors in undergraduates. A successful program for at-risk students will also profoundly impact their academic performance and goal achievement, as well as their lives beyond university. Our partnership will impact knowledge sharing and student training opportunities. With a diversity of academic and non-academic partners and an integrative knowledge sharing approach, the investigator will share results with many audiences throughout the project. The academic researchers have recognized expertise in training and mentoring students. Further, trainees will be exposed to many opportunities and settings both inside and outside of the university in which to apply their research skills to substance misuse prevention.

DETAILED DESCRIPTION:
The UniVenture program is a wellness program designed for university students, to be tested at 5 university-based sites (Dalhousie University, St. Francis Xavier University, York University, Université de Montréal, and University of British Columbia-Okanagan), and based on an existing, successful, and internationally recognized and -utilized program called PreVenture (designed for high school students). PreVenture is a selective personality-targeted approach based on an etiologic model of substance misuse behaviors, outlined and validated by Drs. Stewart (Project Director [PD]) and Conrod (Co-Applicant [CA]). PreVenture targets personality-specific motivational pathways to substance misuse, AS, HOP, SS, and IMP, each associated with different motives for substance use, substance use profiles, and patterns of emotional distress and risk-taking. Well-controlled studies show PreVenture reduces or delays teens' binge drinking, illicit drug use, and associated emotional problems by 30-80% with effects lasting at least 2 years. While PreVenture: (a) was designed for and is effective for high school students, its efficacy in university students is untested; (b) is effective for alcohol and cannabis use, its effects on prescription drug misuse are unknown; and (c) works to reduce student distress, it is untested for preventing academic struggles and university drop out. These latter academic outcomes are of major concern to our Student Affairs partners given the current shockingly high university drop-out rates (18.7-36.9%) and strong ties of student substance misuse and distress with poorer academic outcomes. The purpose of the UniVenture study is to measure the efficacy the developmentally adapted program has on primary outcomes of (1) Reduction of alcohol-related harms in undergraduates (2) Reduction of cannabis-related harms in undergraduates (3) Changes in the student wellbeing in undergraduates. Secondary outcomes are (1) Differences in semester GPA between treatment groups. (2) Changes in scores on the undergraduates' Academic retention measure (3) Changes in scores on the undergraduates' Academic challenges measure (4) Changes in scores on the undergraduate self-regulated learning (SRL) behaviour measure and Self-efficacy beliefs for undergraduates' success measures (5) Reduction in score of hazardous drinkers in undergraduates.

Barriers to accessing evidence-based programs contribute to the ineffectiveness of campus-based substance misuse prevention. These barriers include students' time commitments, lack of available services, fear of stigma, and long wait lists which may discourage students from seeking or engaging in existing programs, leading to more severe problems before participants receive help. A distance-delivery approach involves using remote communication technologies (e.g., web-based, email, chat) to link students with a facilitator in place of face-to-face meetings. This may improve access for those with difficulties getting to services or increase confidentiality through engagement from a private location. The investigator proposes a novel randomized controlled study to test the relative effects of our personality-targeted wellness program on hazardous drinking, cannabis use, and uptake of prescription drug misuse among high-personality-risk 1st and 2nd year undergraduates and delivered in 2 formats: traditional face-to-face vs. an innovative and more accessible technology-assisted distance-delivery by well-trained and supervised program facilitators. These two active program conditions will be compared to a services-as-usual only control condition to evaluate how this program compares to what Student Affairs unit partners already do. Withholding the program from at-risk undergraduates randomized to the services-as-usual only control group might be seen as problematic; however, the program's efficacy is untested at the emerging adulthood (EA) developmental stage and in the university context. If the distance-delivered program is shown effective, control condition participants will be sent a free link to the relevant personality-matched web-based materials after the 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1st and 2nd year undergraduate students (either part-time or full-time enrollment)
* Age between 18- 25 years
* Have used alcohol and/or cannabis and/or any other substance in the past 3 months,
* Score at least 0.5 standard deviation (SD) above the population-specific norm on 1 of 4 personality traits on the Substance Use Risk Profile Scale (SURPS) (i) Anxiety Sensitivity (AS) (ii) Hopelessness (HOP) (iii) Sensation Seeking (SS) and (iv) Impulsive (IMP)

Exclusion Criteria:

• Unwilling to participate

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-11 (Actual); Primary Completion 2024-02-08 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in alcohol-related harms in undergraduates | Past 3 months
  Alcohol use as a continuous measure of alcohol-related harm. The Brief-Young Adult Alcohol Consequences Questionnaire (B-YAACQ) is a 24-item scale that will be used to measure changes in the experiences of alcohol-related harms in the past 3 months. The response options include (1) Yes, in the past 3 months, (2) Yes, but not in the past 3 months (3) No. This measure will be scored as the number of adverse consequences experienced in the last three months on a continuous scale from 0-24.
  [Higher scores indicate greater adverse alcohol consequences]
Changes in cannabis-related harms in undergraduates | Past 3 months
  Cannabis use as a continuous measure of cannabis-related harm. The Brief Marijuana Consequences Questionnaire (BMACQ) is a 21-item scale that will be used to measure changes in participants' reported experiences of cannabis-related harms in the past 3 months. The response options include (1) Yes, in the past 3 months, (2) Yes, but not in the past 3 months (3) No. This measure will be scored as the number of adverse consequences experienced in the last three months on a continuous scale from 0-21.
  [Higher scores indicate greater adverse cannabis consequences]
Changes in the student wellbeing in undergraduates | Past 3 months
  It will be measured by the Patient Health Questionnaire Anxiety-Depression Scale (PHQ-ADS) - which combines the Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder (GAD-7) scales - as a composite measure of depression and anxiety. Response option of Generalized Anxiety Disorder (GAD-7) is (1) Not at all (2) Several days (3) More than half of the days (4) Nearly every day. Response option of Patient Health Questionnaire (PHQ-9) is (1) Not at all (2) Several days (3) Over half the days (4) Nearly every day.
  [Higher scores indicate higher mental wellbeing]

SECONDARY OUTCOMES:
Differences in semester GPA between treatment groups. | Through study completion, an average of 1 year
  Semester-wise grade point average [GPA] as a proxy of Undergraduates' academic performance (i.e., objective indices of grades). GPA data retrieved from the registrar's office at each site will be converted to a common 6-point GPA scale since different university sites use different GPA scales (%, 5-point GPA, 9-point GPA). The scale ranges from 1 to 6 where 1 indicates lower performance and 6 indicates higher performance.
  [Higher scores indicate higher GPA in that semester.]
Changes in scores on the undergraduates' Academic retention measure | Through study completion, an average of 1 year
  Measured by the 6-item self-reported Academic outcome survey: Academic experience scale. Item response options include (1) Strongly disagree (2) Disagree (3) Neither agree nor disagree (4) Agree (5) Strongly agree. A total score is derived by summing scores across the 6 items.
  [Higher scores indicate higher academic retention].
Changes in scores on the undergraduates' Academic challenges measure | Past 2 weeks
  This is assessed with a 35-item Academic outcome survey. This composite score [Self-Regulated Learning -Challenges Scale (SRL-C)] will represent the academic challenges experienced. Item response options range from: (1) Strongly disagree to (5) Strongly agree.
  The composite score is comprised of five areas of academic challenges typically reported by undergraduate students: (1) Motivation (e.g., challenges initiating and sustaining engagement); (2) Goal and time management (e.g., challenges making deadlines, or managing priorities) (3) Cognitive (challenges maintaining focus, understanding course material (4) Socio-emotional (challenges adjusting to new academic expectations; balancing health and well-being); and (5) Meta-cognitive (challenges setting goals or choosing strategies).
  [Higher scores on the composite indicate greater levels of academic challenges being experienced by the student.]
Changes in scores on the undergraduate self-regulated learning (SRL) behaviour measure and Self-efficacy beliefs for undergraduates' success measures | Past 2 weeks
  Two separate scales [SRL Self-Regulated Learning -Practices Scale (SRL-P) and Self-Regulated Learning -Challenges Scale (SRL-C)] will be combined and consist of 35 items from the Academic outcome survey with response options of (1) Strongly disagree (2) Disagree (3) Neutral (4) Agree (5) Strongly agree.
  [Higher scores indicate more proactive self-regulated learning behaviours/practices and indicate stronger belief about academic success]
Changes in score of hazardous drinkers in undergraduates | Past 3 months
  This 3-item The Alcohol Use Disorders Identification Test Consumption screening tool (AUDIT-C) questions (composite score) capture individuals who are hazardous drinkers or who have alcohol use disorders (including alcohol abuse or dependence). It is scored on a scale of 0-12 points (each item has maximum of 4 score where 0 reflect no alcohol use). In men, a score of 4 points or more is considered positive for alcohol misuse; in women, a score of 3 points or more is considered positive.
  Generally, the higher the AUDIT-C score, the higher the likelihood of affecting health and safety due to individual's drinking.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry H Stewart, Study Director — Dalhousie University; Patricia Conrod, Principal Investigator — Université de Montréal; Kara Thompson, Principal Investigator — St. Francis Xavier University; Matthew T Keough, Principal Investigator — York University; Marvin Krank, Principal Investigator — University of British Columbia- Okanagan; Allyson Hadwin, Principal Investigator — University of Victoria
Locations (5):
- Canada (5):
  - University of British Columbia-Okanagan campus, Kelowna, British Columbia
  - St. Francis Xavier University, Antigonish, Nova Scotia
  - Dalhousie University, Halifax, Nova Scotia
  - York University, Toronto, Ontario
  - Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szalavitz, M. (2016, September 29). The 4 traits that put kids at risk for addiction. The New York Times. Retrieved from https://www.nytimes.com/2016/10/04/well/family/the-4-traits-that-put-kids-at- risk-for-addiction.html
- [Background] Nair, R. (2017, January 22). Vernon, B. C. schools to pilot program that identifies addiction personality traits. CBC News. Retrieved from https://www.cbc.ca/news/canada/british-columbia/vernon-b- c-schools-to-pilot-program-thatidentifies-addiction-personality-traits-1.3942792
- [Background] UNESCO, UNODC, & WHO. (2017). Education sector responses to the use of alcohol, tobacco and drugs. In the UNESCO series Good Policy and Practice in Health Education. Retrieved from http://www.who.int/substance_abuse/activities/education_sector/en/
- [Background] Substance Abuse and Mental Health Services Administration (US); Office of the Surgeon General (US). Facing Addiction in America: The Surgeon General's Report on Alcohol, Drugs, and Health [Internet]. Washington (DC): US Department of Health and Human Services; 2016 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK424857/ PMID 28252892
- [Background] Conrod PJ, Stewart SH, Comeau N, Maclean AM. Efficacy of cognitive-behavioral interventions targeting personality risk factors for youth alcohol misuse. J Clin Child Adolesc Psychol. 2006 Dec;35(4):550-63. doi: 10.1207/s15374424jccp3504_6. PMID 17007600
- [Background] Woicik PA, Stewart SH, Pihl RO, Conrod PJ. The Substance Use Risk Profile Scale: a scale measuring traits linked to reinforcement-specific substance use profiles. Addict Behav. 2009 Dec;34(12):1042-55. doi: 10.1016/j.addbeh.2009.07.001. Epub 2009 Jul 8. PMID 19683400
- [Background] Castellanos-Ryan, N., & Conrod, P. J. (2012). Personality and substance misuse: Evidence for a four-factor model of vulnerability. In Verster, J. C., Brady, K., Galanter, M., & Conrod, P. J. (Eds.), Drug abuse and addiction in medical illness: Causes, consequences and treatment (pp. 47-62). New York: Springer.
- [Background] Stewart, S. H., Grant, V. V., Mackie, C. J., & Conrod, P. J. (2016). Comorbidity of anxiety and depression with substance use disorders. In K. Sher (Ed.), The Oxford Handbook of Substance Use Disorders. New York: Oxford University Press.
- [Background] Conrod PJ, Pihl RO, Stewart SH, Dongier M. Validation of a system of classifying female substance abusers on the basis of personality and motivational risk factors for substance abuse. Psychol Addict Behav. 2000 Sep;14(3):243-56. doi: 10.1037//0893-164x.14.3.243. PMID 10998950
- [Background] Conrod PJ, Castellanos N, Mackie C. Personality-targeted interventions delay the growth of adolescent drinking and binge drinking. J Child Psychol Psychiatry. 2008 Feb;49(2):181-90. doi: 10.1111/j.1469-7610.2007.01826.x. PMID 18211277
- [Background] Conrod PJ, Castellanos-Ryan N, Strang J. Brief, personality-targeted coping skills interventions and survival as a non-drug user over a 2-year period during adolescence. Arch Gen Psychiatry. 2010 Jan;67(1):85-93. doi: 10.1001/archgenpsychiatry.2009.173. PMID 20048226
- [Background] O'Leary-Barrett M, Mackie CJ, Castellanos-Ryan N, Al-Khudhairy N, Conrod PJ. Personality-targeted interventions delay uptake of drinking and decrease risk of alcohol-related problems when delivered by teachers. J Am Acad Child Adolesc Psychiatry. 2010 Sep;49(9):954-963.e1. doi: 10.1016/j.jaac.2010.04.011. Epub 2010 Jul 31. PMID 20732631
- [Background] Castellanos, N., & Conrod, P. J. (2006). Brief interventions targeting personality risk factors for adolescent substance misuse reduce depression, panic, and risk-taking behaviors. Journal of Mental Health, 15, 645-658.
- [Background] Mahu IT, Doucet C, O'Leary-Barrett M, Conrod PJ. Can cannabis use be prevented by targeting personality risk in schools? Twenty-four-month outcome of the adventure trial on cannabis use: a cluster-randomized controlled trial. Addiction. 2015 Oct;110(10):1625-33. doi: 10.1111/add.12991. Epub 2015 Jul 14. PMID 26011508
- [Background] MacLean's magazine (January 8, 2018). Canadian universities with the highest (and lowest) graduation rates. Retrieved from https://www.macleans.ca/education/canadian-universities-with-the- highest-and-lowest-graduation-rates/
- [Background] Thombs DL, Olds RS, Bondy SJ, Winchell J, Baliunas D, Rehm J. Undergraduate drinking and academic performance: a prospective investigation with objective measures. J Stud Alcohol Drugs. 2009 Sep;70(5):776-85. doi: 10.15288/jsad.2009.70.776. PMID 19737503
- [Background] Dyson R, Renk K. Freshmen adaptation to university life: depressive symptoms, stress, and coping. J Clin Psychol. 2006 Oct;62(10):1231-44. doi: 10.1002/jclp.20295. PMID 16810671
- [Background] Olthuis, J. V., Watt, M. C., & Stewart, S. H. (2013). Increasing access to evidence-based interventions: The role of technology. Psynopsis, Summer.